CLINICAL TRIAL: NCT04928352
Title: Preemptive Nebulized Bupivacaine for Pain Control After Cleft Palate Repair in Children: A Randomized Double Blind Controlled Trial
Brief Title: Nebulized Bupivacaine Analgesia for Cleft Palate Repair
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300615
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Experimental): Nebulized Bupivacaine 0.50% 0.50 mg.kg-1
  Interventions: Drug: Bupivacaine Hydrochloride
- Group C (Placebo Comparator): Same volume of nebulized saline placebo
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Preoperative Nebulized Bupivacaine 0.50% 0.50 mg.kg-1
  Other Names: marcaine
  Arms: Group B
Other: 0.9% saline — Preoperative nebulized same volume of saline placebo
  Other Names: Normal saline
  Arms: Group C

SUMMARY:
In this study we introduce a potent local anesthetic; bupivacaine 0.5% in 0.5 mg/kg dose by nebulization as a preemptive analgesia to compare efficacy and safety in children with cleft palate repair.

DETAILED DESCRIPTION:
A written informed consent will be taken from the guardian of children. Patients will be assigned randomly to two groups (30 subjects each) to be anesthetized. The study drug will be delivered in opaque bags labeled "study drug" and 60 patients will be allocated in two groups (of 30 patients each) to receive; Nebulized plain Bupivacaine 0.50% 0.50 mg.kg-1 (Group B) or same volume of saline placebo (Group C).

ELIGIBILITY:
Inclusion Criteria:

* Children (age 1-7 years) of American Society of Anaesthesiologists physical status (ASA) I-II
* Elective cleft palate repair ± cleft lip surgery under general anesthesia .

Exclusion Criteria:

* Coronary artery disease
* Hypertension
* Developmental delay
* Allergy to study drug

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
the total postoperative consumption of rescue analgesics | 24 hour after surgery
  Patients will receive IV paracetamol 15 mg.kg-1 as rescue analgesia if requested and if FLACC scores were ≥4. The FLACC (Face, Legs, Activity, Cry, Consolability). We rate the child in each of the five measurement categories, add together, and document total pain score (0 - 10) where 0= relaxed and no pain, 1-3= mild pain/discomfort, 4-6= moderate pain, 7-10= severe discomfort/pain. The scale will be recorded on admission to PACU (baseline), and at 30 minutes, 1, 3, 6, 12 and 24 hour postoperative.

SECONDARY OUTCOMES:
Postoperative FLACC score | 24 hour postoperative
  The FLACC (Face, Legs, Activity, Cry, Consolability) is a behavioural pain assessment scale for use in non-verbal or pre-verbal patients unable to self-report their level of pain.We rate the child in each of the five measurement categories, add together, and document total pain score (0 - 10) where 0= relaxed and no pain, 1-3= mild pain/discomfort, 4-6= moderate pain, 7-10= severe discomfort/pain. The scale will be recorded on admission to PACU (baseline), and at 30 minutes, 1, 3, 6, 12 and 24 hour postoperative.
The time to first request for rescue analgesics | 24 hour postoperative
  Recording the first time when patients will receive IV paracetamol 15 mg.kg-1 as rescue analgesia if requested and if FLACC scores were ≥4.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chiono J, Raux O, Bringuier S, Sola C, Bigorre M, Capdevila X, Dadure C. Bilateral suprazygomatic maxillary nerve block for cleft palate repair in children: a prospective, randomized, double-blind study versus placebo. Anesthesiology. 2014 Jun;120(6):1362-9. doi: 10.1097/ALN.0000000000000171. PMID 24525630